CLINICAL TRIAL: NCT07071558
Title: A Phase 1, Parallel, Randomized, Multi-center Study to Evaluate the Safety and Immunogenicity of Different LNP Formulations of mRNA Vaccines Using the RSV Monovalent Antigen in Healthy Participants 18 to 49 Years of Age
Brief Title: Study to Evaluate the Safety and Immunogenicity of Investigational Vaccines Using the RSV (Respiratory Syncytial Virus) Monovalent Antigen in Healthy Participants 18 to 49 Years of Age
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00026; WHO UTN (Other: U1111-1321-1812)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus Immunization
Keywords: RSV; RSV Infection; RSV Vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators, study site staff, laboratory personnel, outcome assessors, and participants will be blinded throughout the study. Study staff preparing and administering the study interventions will be unblinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- RSV Formulation 1 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 1 dose
- RSV Formulation 2 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 2 dose
- RSV Formulation 3 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 3 dose
- RSV Formulation 4 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 4 dose
- RSV Formulation 5 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 5 dose
- RSV Formulation 6 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 6 dose
- Control group 1 dose 1 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 7 dose
- Control group 2 dose 2 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV vaccines according to their randomization schedule.
  Interventions: Biological: RSV vaccine formulation 8 dose

INTERVENTIONS:
Biological: RSV vaccine formulation 1 dose — Suspension for injection. Route of administration: IM injection
  Arms: RSV Formulation 1
Biological: RSV vaccine formulation 2 dose — Suspension for injection. Route of administration: IM injection
  Arms: RSV Formulation 2
Biological: RSV vaccine formulation 3 dose — Suspension for injection. Route of administration: IM injection
  Arms: RSV Formulation 3
Biological: RSV vaccine formulation 4 dose — Suspension for injection. Route of administration: IM injection
  Arms: RSV Formulation 4
Biological: RSV vaccine formulation 5 dose — Suspension for injection. Route of administration: IM injection
  Arms: RSV Formulation 5
Biological: RSV vaccine formulation 6 dose — Suspension for injection. Route of administration: IM injection
  Arms: RSV Formulation 6
Biological: RSV vaccine formulation 7 dose — Suspension for injection. Route of administration: IM injection
  Arms: Control group 1 dose 1
Biological: RSV vaccine formulation 8 dose — Suspension for injection. Route of administration: IM injection
  Arms: Control group 2 dose 2

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of different liponanaoparticle (LNP) formulations of modified ribonucleic acid (mRNA) vaccines using the RSV pre-F antigen in healthy participants 18 to 49 years of age.

-Each participant will remain in the study for approximately 6 months.

* The study intervention will be administered as a single intramuscular (IM) dose in the upper arm on Day 1 (D01).
* The visit frequency will include 1 Screening Visit, 4 planned site visits to occur on D01, D03, D08, and D29, and 2 telephone calls to occur at Month (M)3 and M6.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 49 years on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and of the following conditions applies:

  * Is of NCBP (Non-Child-Bearing Potential). To be considered of NCBP, a female must be post-menopausal for at least 1 year, or surgically sterile. OR
  * Is of CBP (Child-Bearing Potential) and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Presence of any unsolicited systemic adverse events (aes) | Within 30 minutes after each vaccine injection
  Number of participants experiencing immediate AEs
Presence of solicited injection site reactions (ie, pre-listed in the participant's diary and in the eCRF (electronic case report form) | Through 7 days after each vaccine injection
  Number of participants experiencing solicited injection site reactions
Presence of solicited systemic reactions (ie, pre-listed in the participant diary and in the CRF) | Through 7 days after each vaccine injection
  Number of participants experiencing solicited systemic reactions
Presence of unsolicited AEs | Day 1 through day 29
  Number of participants experiencing unsolicited AEs
Presence of SAEs (Serious Adverse Events) and AESIs (Adverse Events of Special Interest) | Throughout study, approximately 6 months
  Number of participants experiencing SAEs and AESIs
Presence of out-of-range biological test results (including shift from baseline values) | Through 7 days after each vaccine injection
  number of participants with out-of-range biological tests
RSV A nAb (Neutralizing Antibodies) titers | At day 1 and day 29

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Site # 0361003, Wollongong, New South Wales
  - Site # 0361006, Brisbane, Queensland
  - Site # 0361005, Morayfield, Queensland
  - Site # 0361004, Southport, Queensland
  - Site # 0361002, Bayswater, Victoria
  - Site # 0361001, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26837&tenant=MT_SNY_9011